CLINICAL TRIAL: NCT00800345
Title: A Phase I Trial of Oral Metronomic Topotecan in Combination With Oral Pazopanib Utilizing a Daily Dosing Schedule to Treat Recurrent or Persistent Gynecologic Tumors
Brief Title: Phase I Trial of Oral Metronomic Topotecan and Oral Pazopanib to Treat Recurrent/Persistent Gynecologic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vector Oncology (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATDTRPST0802
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2016-12

CONDITIONS: Gynecologic Tumors
Keywords: Gynecologic tumors
MeSH Terms: interventions — Topotecan; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimenal (Experimental): Metronomic oral topotecan and oral pazopanib will be administered by mouth beginning on Cycle 1 Day 1. Patients will be enrolled and observed for dose limiting toxicity (DLT) for 1 cycle of treatment. Dose modification of the combination will depend on the number of patients experiencing DLT(s) at each dose level.
  Interventions: Drug: Oral Topotecan; Drug: Pazopanib

INTERVENTIONS:
Drug: Oral Topotecan — Starting on Cycle 1 Day 1, each subject will receive the assigned dose of topotecan administered by mouth.
  Other Names: Hycamtin capsules
Drug: Pazopanib — Starting on Cycle 1 Day 1, each subject will receive the assigned dose of pazopanib administered by mouth.
  Other Names: GW786034; Votrient

SUMMARY:
This is a Phase 1, dose-escalation study in female patients with recurrent or persistent gynecologic tumors.

DETAILED DESCRIPTION:
This is a Phase 1, dose-escalation study in female patients with recurrent or persistent gynecologic tumors. The study will include a Screening Phase, a Treatment Phase and a Followup Phase. In the Screening Phase the subject's eligibility for study participation will be determined; this phase can last up to 28 days. The Treatment Phase will begin when the subject starts study treatment and will continue until the subject is removed from study treatment. The Follow-up Phase will last for 30 days after the subject ends study treatment. The study will be conducted at approximately 1 site. Treatment cycle length is 28 days. Radiologic imaging will be repeated after every 2 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to the performance of study specific procedures, and must be willing to comply with treatment and follow-up.
* Female patients, greater than 18 years of age with a histologically confirmed recurrent/persistent gynecologic malignancy.
* For patients with recurrent/persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma: persistent disease = progression during primary platinum therapy; recurrent disease = disease that recurs ≤ 12 months after discontinuing primary platinum therapy; if disease recurrence occurs > 12 months after discontinuing primary platinum therapy, there must be progression either during a 2nd platinum therapy or < 6 months after discontinuing the 2nd platinum therapy.
* For patients with other gynecologic malignancies:

  * Malignancy is metastatic or unresectable and no curative or palliative measures exist or are no longer effective.
  * Maximum of two total prior treatments (this includes neoadjuvant, adjuvant, and metastatic settings) for the recurrent or persistent gynecologic tumors including chemotherapy, hormonal therapy, investigational therapy, radiation therapy, etc.)
* Disease may be measurable or non-measurable according to RECIST version 1.0
* Gynecologic Oncology Group (GOG) performance status of 0,1,or 2
* Must have a life expectancy of at least six months
* Adequate bone marrow, liver, renal, and cardiac function at study entry as assessed by the following:

  * Hemoglobin > 9.0 g/dL.
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
  * Platelet count ≥ 100 x 10^9/L.
  * Prothrombin time (PT) or international normalized ratio (INR) < 1.2 x upper limit of normal (ULN).
  * Partial thromboplastin time (PTT) < 1.2 x ULN.
  * Total bilirubin ≤ 1.5 x ULN.
  * Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN.
  * Creatinine ≤ 1.5 mg/dL or if serum creatinine is greater than 1.5 mg/dL, calculated creatinine clearance must be > 50 mL/min
  * Urine dipstick for protein < 2+ or urine protein creatinine (UPC) ratio < 1.0.
  * Left ventricular ejection fraction (LVEF) ≥ 50% or the institutional lower limit of normal (LLN)
* Patients must be physiologically incapable of becoming pregnant, be postmenopausal, or have a negative pregnancy test and agree to use adequate contraception.

Exclusion Criteria:

* Treatment naive patients.
* Repetitive or prolonged neutropenia or thrombocytopenia during previous therapy.
* Concurrent malignancy other than malignancies under study. Subjects who have had another malignancy and have been disease free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* Prior radiation therapy.
* Myelosuppressive chemotherapy within the past 28 days or has not recovered from the myelosuppressive effects of recent chemotherapy.
* Use of an investigational agent, including an investigational anti-cancer agent, immunotherapy, biological therapy, or hormonal therapy within 28 days prior to the first dose of study treatment.
* Prior major surgery or trauma within 28 days prior to the first dose of study treatment and/or presence of any non-healing wound, fracture, or ulcer.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis.
* Inability to swallow a capsule or clinically significant gastrointestinal abnormalities including, but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel that could affect the absorption of study treatment
  * Active peptic ulcer disease
  * Inflammatory bowel disease
  * Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
  * Unresolved bowel obstruction or diarrhea ≥ Grade 1
  * Known intraluminal metastatic lesion(s) with risk of bleeding
* Known endobronchial lesions or involvement of large pulmonary vessels by tumor.
* Presence of uncontrolled infection.
* Prolongation of corrected QT interval > 480 milliseconds.
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension (defined as systolic blood pressure of > 140 mmHg or diastolic blood pressure of > 90 mmHg). Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.
* History of cerebrovascular accident, transient ischemic attack, pulmonary embolism, or insufficiently treated deep vein thrombosis (DVT) within the past 6 months. Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
* Evidence of active bleeding or bleeding diathesis.
* Recent hemoptysis in excess of 2.5 mL within 8 weeks of 1st dose of study treatment.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Use of any prohibited medication within 14 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study treatment and during the study.
* Prior use of any investigational or licensed anti-angiogenic agent, including topotecan, bevacizumab, thalidomide, and agents that target vascular endothelial growth factor (VEGF), VEGF receptors, or platelet-derived growth factor (PDGF).
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity, except alopecia.
* Known hypersensitivity to topoisomerase I inhibitors or pazopanib.
* Administration of any non-oncologic investigational drug within 30 days or five half-lives of a drug (whichever is longer) prior to the first dose of study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-04; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Tillmanns, MD, Principal Investigator — The West Clinic
Locations (1):
- The West Clinic, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Metronomic oral topotecan and oral pazopanib will be administered by mouth beginning on Cycle 1 Day 1. Patients will be enrolled and observed for dose limiting toxicity (DLT) for 1 cycle of treatment. Dose modification of the combination will depend on the number of patients experiencing DLT(s) at each dose level.
  Oral Topotecan: Starting on Cycle 1 Day 1, each subject will receive the assigned dose of topotecan administered by mouth.
  Pazopanib: Starting on Cycle 1 Day 1, each subject will receive the assigned dose of pazopanib administered by mouth.
Period: Overall Study
Arm/Group | Experimental
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.88 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Time Frame: Cycle 1 (28 days)
Measure: Number; unit: participants
Arm/Group | Experimental
Number analyzed (Participants) | 33
participants
  Experienced a DLT | 8
  Did not experience a DLT | 23
  Unevaluable | 2

2. Secondary Outcome: Treatment Response
Description: Treatment response was evaluated using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter (LD) of target lesions; Stable Disease (SD) is neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; Progressive Disease (PD) is the increase in existing lesions or new lesions.
Time Frame: After every 2 cycles of treatment beginning on Cycle 1 Day 1, up to 38 months
Measure: Number; unit: participants
Arm/Group | Experimental
Number analyzed (Participants) | 33
participants
  Complete Response | 4
  Partial Response | 5
  Stable Disease | 13
  Progressive Disease | 10
  Not Evaluable | 1

ADVERSE EVENTS:
Arm/Group | Experimental
Serious Adverse Events (participants affected / at risk) | 11/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=33)
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=33)
Anaemia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 2
Hypoacusis (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Ocular hyperaemia (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 20
Dyspepsia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 5
Gastrointestinal fistula (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 23
Oral disorder (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 8
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 18
Catheter site pain (General disorders) | 1
Chest discomfort (Hepatobiliary disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 20
Influenza like illness (General disorders) | 1
Mucosal inflammation (General disorders) | 2
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 3
Tenderness (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Allergy to arthropod sting (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 2
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 12
Vulvovaginal mycotic infection (Infections and infestations) | 1
Administration related reaction (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Lipase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 10
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Anosmia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 18
Headache (Nervous system disorders) | 8
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 10
Urinary tract disorder (Renal and urinary disorders) | 2
Female genital tract fistula (Reproductive system and breast disorders) | 1
Hydrometra (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Vaginal fistula (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythemas (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Skin mass (Skin and subcutaneous tissue disorders) | 1
Sinus operation (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 5
Lymphoedema (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less